CLINICAL TRIAL: NCT04374747
Title: Fruit and Vegetable Intervention in Lactating Women to Reduce Breast Cancer Risk: Effects on Breast Cell DNA Methylation, Breast Inflammation,and Weight
Brief Title: Fruit and Vegetable Intervention in Lactating Women to Reduce Breast Cancer Risk
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Massachusetts, Amherst (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2019-5382; 1R01CA230478-01A1 (NIH)
Record Dates: First submitted 2020-04-30; First posted 2020-05-05 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-04

CONDITIONS: Breast Cancer Female; Inflammation; Postpartum Weight Retention; Diet, Healthy; Risk Reduction
MeSH Terms: conditions — Inflammation; Gestational Weight Gain; Risk Reduction Behavior | interventions — Nutrition Assessment

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Key laboratory analyses will conducted by laboratories blinded to intervention arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dietary Intervention (Experimental): Intensive dietary counseling and fruit and vegetable box delivery.
  Interventions: Behavioral: Dietary Counseling
- Information (No Intervention): Control condition of information on healthy eating during breastfeeding

INTERVENTIONS:
Behavioral: Dietary Counseling — The counseling approach will employ strategies shown to be successful in previous and ongoing dietary modification studies including supportive and motivational interviewing techniques. Each woman in the diet intervention group will be assigned a trained nutrition coach/counselor. Counselors will focus on helping participants identify and address barriers to achieving the goal of consuming at least 8 to 10 servings of nutrient dense fruits and vegetables each day (e.g., modifying recipes and food preparation). Participants will also receive weekly boxes of fruits and vegetables .
  Arms: Dietary Intervention

SUMMARY:
Mechanistic data show that compounds in fruits and vegetables have anti-inflammatory and anti-carcinogenic properties that can reduce breast cancer risk. However, observational and interventional studies have provided mixed results, and a recent report by the American Institute for Cancer Research (AICR) concludes that the data are insufficient but suggestive that non-starchy vegetables and foods containing carotenoids reduce risk. Measurement error, relatively low levels of carotenoid-rich fruit and vegetable intake in the study populations, emphasis on diet in later adulthood, and confounding factors likely contribute to the weak associations. Therefore, the investigators will conduct a randomized diet intervention trial in young women to assess the extent to which at least 8 to 10 daily servings of deeply pigmented and nutrient dense fruits and vegetables reduces biomarkers of breast cancer risk. The intervention is focused on breastfeeding women because: 1) pregnancy and lactation are normal early life course events; 2) the risk of pregnancy-associated breast cancer (PABC) is increased for up to 10 years postpartum; 3) a dietary intervention to reverse the detrimental molecular changes associated with puberty and pregnancy is more likely to be successful in younger than in older women;4) a diet rich in fruits and vegetables is hypothesized to reduce the inflammation during lactation/weaning and lower PABC risk; 5) postpartum lactating women may be a highly motivated population; and 6) breastmilk provides access to the breast microenvironment and breast epithelial cells to non-invasively assess the diet intervention directly in the breast. Four hundred nursing mothers will be randomly assigned to either the intervention arm, in which they are asked to increase fruit and vegetable intake to at least 8 to 10 daily servings for one year, or to a control condition in which participants receive a dietary guideline for breastfeeding mothers. Women in the intervention arm will receive counseling and boxes of fruits and vegetables for the first 20 weeks, after which they will continue to receive counseling. Changes in DNA methylation and cytokine profiles in breastmilk will be evaluated. Maternal weight and body fat distribution, and infant growth will be monitored. These results will greatly expand our knowledge of how diet alters molecular pathways in a specific organ, ultimately contributing to both breast cancer etiology and prevention.

DETAILED DESCRIPTION:
Overview of home visits and activities completed by all participants

Visit 1 Introductory Visit (1.5 hours) 24-Hour Dietary Recalls completed during the week (1-2 hours) Occurs at 5 weeks postpartum

* Informed Consent document administered.
* Public Data Sharing Informed Consent document administered.
* Three questionnaires: New Moms Health, Physical Activity, and Breastfeeding Practices
* Maternal height, weight, and waist circumference measured.
* Instructions provided for future collection of biospecimens.
* Complete one 24-Hour Dietary Recall
* Instructions provided for two additional 24-Hour Dietary Recalls.

Visit 2 Sample Collection 1 (1.5 hours) Occurs at 6 weeks postpartum

* Provide bilateral breast milk samples and completed questionnaire.
* Provide infant stool sample and completed questionnaire.
* Two questionnaires: Infant Feeding, and Medication & Supplement
* Infant length and weight measured.
* Maternal and infant skin carotenoids measured.
* Nutrition education provided.
* Optional collection of maternal stool sample and completed questionnaire.

Visit 3 Sample Collection 2 (1.5 hours) 24-Hour Dietary Recalls completed during the week (1-2 hours) Occurs at 16 weeks postpartum

* Provide bilateral breast milk samples and completed questionnaire.
* Provide infant stool sample and completed questionnaire.
* Three questionnaires: Physical Activity, Infant Feeding, and Medication & Supplement
* Infant length and weight measured.
* Maternal weight and waist circumference measured.
* Maternal and infant skin carotenoids measured.

Visit 4 Sample Collection 3 (1.5 hours) 24-Hour Dietary Recalls completed during the week (1-2 hours) Occurs at 26 weeks postpartum

* Provide bilateral breast milk samples and completed questionnaire.
* Provide infant stool sample and completed questionnaire.
* Three questionnaires: Physical Activity, Infant Feeding, and Medication & Supplement.
* Infant length and weight measured.
* Maternal weight and waist circumference measured.
* Maternal and infant skin carotenoids measured.
* Optional collection of maternal stool samples and completed questionnaire.

Visit 5 Sample Collection 4 (1.5 hours) 24-Hour Dietary Recalls completed during the week (1-2 hours) Occurs at 58 weeks postpartum

* Provide bilateral breast milk samples and completed questionnaire.
* Provide infant stool sample and completed questionnaire.
* Four questionnaires: Physical Activity, Infant Feeding, Medication and Supplement, and Breast Health
* Infant length and weight measured.
* Maternal weight and waist circumference measured.
* Maternal and infant skin carotenoids measured.
* Optional collection of maternal stool samples and completed questionnaire.

Annual Follow-up Visit (Maximum of 2) (1 hour) 24-Hour Dietary Recalls completed during the week (1-2 hours) Occurs at one-year intervals after Visit 5

* Three questionnaires: Physical Activity, Breast Health, Young Child Feeding
* Infant height and weight measured.
* Maternal weight and waist circumference measured.
* Maternal and infant skin carotenoids measured.

Monthly Inquiry (1 - 2 minutes) Occurs monthly until no longer breastfeeding

• Complete the Breast Feeding Update Questionnaire online via a survey sent through REDCap, or through a phone call.

ELIGIBILITY:
Inclusion Criteria:

* Have given birth in past five weeks or are currently pregnant
* Breastfeeding baby at entry into the study
* Consuming five or fewer servings of fruits and vegetables daily at baseline
* Live within 25 miles of Amherst MA

Exclusion Criteria:

* Invasive breast cancer
* Any cancer except non-melanoma skin cancer in past five years
* History of Crohn's disease, celiac sprue, or other malabsorption syndrome, which may interfere with digesting or absorption of nutrients
* A personal history of diabetes (excluding gestational diabetes)
* Baseline BMI of <18.5
* Dietary restrictions that prevent participant from eating 8 to 10 servings of fruits and vegetables

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2019-10-24 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
DNA methylation | 20 weeks
  % methylation in 300,000 CpG sites in DNA from sloughed breast epithelial cells from milk
Inflammatory markers in milk | 20 weeks
  Adiponectin, CRP, IFN-y, IL1-beta, Leptin, IL-6, IL-8, TNF-alpha, b-FGF, FLT-1, PLGF, VegF-D
Early weight | 20 weeks
  maternal weight
Early waist circumference | 20 weeks
  maternal waist circumference
One-year Weight | One-year
  maternal weight
One-year Waist Circumference | one year
  maternal weight circumference

OTHER OUTCOMES:
Fruit and Vegetable Intake | one year
  servings per day

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Arcaro, PhD, Principal Investigator — University of Massachusetts, Amherst; Lindiwe Sibeko, PhD, Principal Investigator — University of Massachusetts, Amherst; Susan Sturgeon, DrPH, Principal Investigator — University of Massachusetts, Amherst
Locations (1):
- University of Massachusetts Amherst, Amherst, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to make IPD available to other researchers.

REFERENCES:
- [Background] Essa AR, Browne EP, Punska EC, Perkins K, Boudreau E, Wiggins H, Anderton DL, Sibeko L, Sturgeon SR, Arcaro KF. Dietary Intervention to Increase Fruit and Vegetable Consumption in Breastfeeding Women: A Pilot Randomized Trial Measuring Inflammatory Markers in Breast Milk. J Acad Nutr Diet. 2018 Dec;118(12):2287-2295. doi: 10.1016/j.jand.2018.06.015. Epub 2018 Sep 10. PMID 30213617
- [Derived] Sturgeon SR, Sibeko L, Balasubramanian R, Arcaro KF. New Moms Wellness Study: the randomized controlled trial study protocol for an intervention study to increase fruit and vegetable intake and lower breast cancer risk through weekly counseling and supplemental fruit and vegetable box delivery in breastfeeding women. BMC Womens Health. 2022 Sep 24;22(1):389. doi: 10.1186/s12905-022-01967-9. PMID 36153518